CLINICAL TRIAL: NCT04898777
Title: Endoscopic Ultrasound-Guided Choledochoduodenostomy Versus Endoscopic Retrograde Cholangiopancreatography for Primary Biliary Decompression in Distal Malignant Biliary Obstruction
Brief Title: EUS-Guided Choledochoduodenostomy Versus ERCP for Primary Biliary Decompression in Distal Malignant Biliary Obstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MD.21.03.437
Record Dates: First submitted 2021-05-05; First posted 2021-05-24 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2023-10

CONDITIONS: Malignant Biliary Obstruction
Keywords: ERCP; EUS; Distal Malignant Biliary Obstruction; Choledochoduodenostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ERCP-BD (Active Comparator): ERCP Biliary Drainage by papillary approach with stent placement.
  Interventions: Procedure: Biliary drainage
- EUS-BD (Active Comparator): Endoscopic Ultrasound guided Biliary Drainage by Choledochoduodenostomy with transmural stent placement.
  Interventions: Procedure: Biliary drainage

INTERVENTIONS:
Procedure: Biliary drainage — Biliary decompression in cases of distal malignant obstruction by stent placement either using ERCP or EUS.
  Other Names: Biliary Decompression

SUMMARY:
Malignant biliary obstruction commonly caused by pancreatic adenocarcinoma, cholangiocarcinoma and other etiologies like gallbladder carcinoma, hepatocellular carcinoma, lymphoma, and metastasis to regional solid organs and lymph nodes.

Pancreatobiliary cancers generally present with jaundice, weight loss, and anorexia with significant impact on quality of life, morbidity, and mortality.

The primary goal of diagnosis and management is curative resection but it's difficult due to local invasion and distant metastases at the time of clinical presentation. Biliary decompression helps to reduce symptoms and improve quality of life in patients with malignant biliary obstruction.

Endoscopically placed stents have become the standard of care for non-surgical biliary drainage due to their minimal invasiveness compared to percutaneous drainage.

The standard treatment of obstructive jaundice has been ERCP with biliary stent placement with high success rate in expert hands and low frequency of adverse events.

Endoscopic ultrasound-guided biliary drainage (EUS-BD) has been increasingly used in patients who underwent failed ERCP. EUS-BD can be performed in several ways, choledochoduodenostomy (CDS), hepaticogastrostomy (HGS), antegrade (AG) procedure, and rendezvous (RV) technique.

DETAILED DESCRIPTION:
This study will be a single center, prospective randomized comparative study that includes 50 patients with distal malignant biliary obstruction including pancreatic head masses, distal cholangiocarcinoma or papillary carcinoma.

All patients with inclusion criteria will be recruited in the study by simple random sampling using sealed envelopes until fulfillment of needed sample size for both EUS-BD arm and ERCP-BD arm.

Study tools:

* Informed consent will be obtained from each participant sharing in the study.
* Throughout history taking, complete general examination and local abdominal examination.
* Laboratory investigations: CBC, Serum creatinine, Liver functions tests (AST, ALT and Serum Albumin), Alkaline phosphatase, Serum bilirubin and INR.
* ERCP-BD by papillary approach and EUS-BD by choledochoduodenostomy with transmural stent placement.
* All procedures will be performed under deep sedation or general anesthesia in the left lateral position.
* Procedural time is recorded.
* Technical success is considered after stent placement (expanded and patent) with good bile flow and drainage.
* Follow up:
* Lab investigations will be requested at 2 days, 2 and 4 weeks, 3 and 6 months after the procedure including:

CBC, S.Cr, S.Bil, AST, ALT, S.Alb, ALP and INR.

- Early adverse events (within 48 hours after procedure) including: Pancreatitis, Cholangitis, Bleeding, Perforation and Peritonitis.

* Late adverse events include stent dysfunction either due to food impaction, tumor ingrowth or stent migration.
* Clinical success is considered at 2 weeks if total bilirubin is less than 50% of baseline and at 4 weeks if total bilirubin is less than 3mg/dL.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years and older.
* Presence of locally advanced or metastatic pancreatic head mass on CT or magnetic resonance imaging of the abdomen
* Absence of duodenal obstruction.
* Elevated liver tests with serum bilirubin at least 3 times above the upper limit of normal (1.2 mg/dL).
* Histologic or cytologic diagnosis of malignancy.
* Accept sharing in the study.

Exclusion Criteria:

* Age younger than 18 years.
* Pregnancy.
* Hilar biliary obstruction (as the main lesion or coexisting with distal obstruction).
* Presence of duodenal obstruction.
* Histologic or cytologic diagnosis of malignancy.
* Patients underwent previous intervention for biliary drainage.
* Previously failed biliary cannulation at ERCP.
* Prior biliary sphincterotomy or stent placement.
* Surgically altered anatomy or inability to access the major duodenal papilla.
* Patients unfit for anesthesia.
* Patients having uncorrectable coagulopathy or thrombocytopenia.
* History of allergy to radiocontrast agents.
* Refuse sharing in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
The rate of adverse events | 6 months
  - Early adverse events (within 48 hours after procedure) including: Pancreatitis, Cholangitis, Bleeding, Perforation and Peritonitis.
  - Late adverse events include stent dysfunction either due to food impaction, tumor ingrowth or stent migration

SECONDARY OUTCOMES:
Rate of technical success | During procedure
  Technical success is considered after successful stent placement.
Rate of clinical success | 4 weeks
  Clinical success is considered at 2 weeks if total bilirubin is less than 50 percent of baseline.
Procedural duration | During procedure
  Procedure time was defined as time from biliary cannulation to stent placement in ERCP group, and time from needle puncture of the dilated bile duct to stent placement in EUS-BD group. In cases of difficult cannulation (defined as failed biliary access within 5 min of attempt), we performed early precut fistulotomy for cannulation by experts without involvement of trainees and duodenal intubation time was not included within procedure time.
Reinterventions | 6 months
  Re-endoscopy in cases of stent migration, occlusion by food or tumor ingrowth.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Gaheen, MSc., Principal Investigator — Mansoura University; Ahmed Y Altonbary, MD, Study Director — Mansoura University; Hazem H Alminshawy, Professor, Study Director — Mansoura University; Ahmed G Deiab, A.Professor, Study Director — Mansoura University; Magdy H Atwa, Professor, Study Chair — Mansoura University
Locations (1):
- Specialized Medical Hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No